CLINICAL TRIAL: NCT03763877
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Trial to Assess the Efficacy and Safety of PXL770 Versus Placebo After 12 Weeks of Treatment in Patients With NAFLD
Brief Title: A Study of the Efficacy and Safety of PXL770 Versus Placebo After 12 Weeks of Treatment in Patients With NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PXL770-004
Record Dates: First submitted 2018-11-28; First posted 2018-12-04 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 2-chloro-3-(1-hydroxy-5,6,7,8-tetrahydronaphthalen-2-yl)-6-oxo-5-phenyl-7H-thieno)(2,3-b)pyridin-4-olate potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): PXL770 Dose 1
  Interventions: Drug: PXL770
- Group 2 (Experimental): PXL770 Dose 2
  Interventions: Drug: PXL770
- Group 3 (Experimental): PXL770 Dose 3
  Interventions: Drug: PXL770
- Group 4 (Placebo Comparator): Placebo oral capsule
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: PXL770 — Oral capsule
  Arms: Group 1; Group 2; Group 3
Drug: Placebo Oral Capsule — Oral capsule
  Arms: Group 4

SUMMARY:
This study will assess the efficacy and safety of 3 doses of PXL770 versus placebo after 12 weeks of treatment.

DETAILED DESCRIPTION:
The study will be performed in patients with Nonalcoholic Fatty Liver Disease. The primary endpoint will be the assessment of the change in the percentage of liver fat mass (assessed by MRI-PDFF).

ELIGIBILITY:
Inclusion Criteria:

* Patients have given written informed consent
* Body mass index (BMI) ≥ 25 to ≤ 50 kg/m²
* For patients with type 2 diabetes mellitus: either naive of glucose lowering drug or under stable oral glucose lowering drug
* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/[min*1.73m²]
* Alanine amino transferase (ALT) > 20 IU/L in females and > 30 IU/L in males
* Hepatic steatosis (MRI-PDFF ≥ 10%)
* Effective contraception for women of child bearing potential

Exclusion Criteria:

* Evidence of another form of liver disease
* Evidence of liver cirrhosis
* Evidence of hepatic impairment
* Positive serologic evidence of current infectious liver disease
* History of excessive alcohol intake
* Acute cardiovascular disease with 24 weeks prior to screening
* Uncontrolled high blood pressure
* Any disease which in the Investigator's opinion which in the Investigator's opinion would exclude the patient from the study
* Use of non-permitted concomitant medication
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Study Site 02, Los Angeles, California
  - Study Site 01, Gainesville, Florida
  - Study Site 11, Ocoee, Florida
  - Study Site 15, Orlando, Florida
  - Study Site 10, Athens, Georgia
  - Study Site 03, Indianapolis, Indiana
  - Study Site 07, Marrero, Louisiana
  - Study Site 05, West Monroe, Louisiana
  - Study Site 08, Berlin, New Jersey
  - Study Site 09, Durham, North Carolina
  - Study Site 13, Rapid City, South Dakota
  - Study Site 06, Arlington, Texas
  - Study Site 04, San Antonio, Texas
  - Study Site 12, San Antonio, Texas
  - Study Site 14, Richmond, Virginia

REFERENCES:
- [Derived] Cusi K, Alkhouri N, Harrison SA, Fouqueray P, Moller DE, Hallakou-Bozec S, Bolze S, Grouin JM, Jeannin Megnien S, Dubourg J, Ratziu V. Efficacy and safety of PXL770, a direct AMP kinase activator, for the treatment of non-alcoholic fatty liver disease (STAMP-NAFLD): a randomised, double-blind, placebo-controlled, phase 2a study. Lancet Gastroenterol Hepatol. 2021 Nov;6(11):889-902. doi: 10.1016/S2468-1253(21)00300-9. Epub 2021 Sep 22. PMID 34560015
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34560015/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for the study at 15 sites in the United States between 29Mar19 and 13Mar20.
Pre-assignment Details: Following a Screening period of maximum 2 weeks, eligible participants entered in a single-blind placebo Run-in period of 4 weeks. This Run-in period was set to reduce any bias regarding placebo effect, to assess patient compliance, and to minimize the possible confounding influence of dietary and activity changes. Only participants who have met all the applicable Inclusion criteria and none of the Exclusion criteria at the end the Run-in period were to be randomized.
Groups:
- Placebo: Placebo: Oral capsule
  Two capsules were taken BID with a glass of water at least 15 minutes before a meal in the morning and in the evening time for 12 weeks
- PXL770 250 mg QD: PXL770 250 mg: Oral capsule Placebo: Oral capsule
  Two capsules were taken BID with a glass of water at least 15 minutes before a meal in the morning and in the evening time for 12 weeks:
  * 1 capsule of PXL770 250 mg + 1 capsule of placebo in the morning
  * 2 capsules of placebo in the evening
- PXL770 250 mg BID: PXL770 250 mg: Oral capsule Placebo: Oral capsule
  Two capsules were taken BID with a glass of water at least 15 minutes before a meal in the morning and in the evening time for 12 weeks:
  * 1 capsule of PXL770 250 mg + 1 capsule of placebo in the morning
  * 1 capsule of PXL770 250 mg + 1 capsule of placebo in the evening
- PXL770 500 mg QD: PXL770 250 mg: Oral capsule Placebo: Oral capsule
  Two capsules were taken BID with a glass of water at least 15 minutes before a meal in the morning and in the evening time for 12 weeks:
  * 2 capsules of PXL770 250 mg
  * 2 capsules of placebo in the evening
Period: Overall Study
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Started (Randomized) | 31 | 30 | 31 | 29
Received at Least 1 Dose of Double-blind Study Treatment | 31 | 30 | 30 | 29
Completed the Double-blind Period | 27 | 26 | 25 | 24
Completed (Completed the follow-up period) | 26 | 26 | 24 | 24
Not Completed | 5 | 4 | 7 | 5
Not completed — Withdrawal by Subject | 3 | 1 | 3 | 4
Not completed — Adverse Event | 1 | 1 | 3 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat set (ITTS), defined as all as-randomized patients who received at least one dose of study treatment.
Groups:
- Placebo; PXL770 250 mg QD; PXL770 250 mg BID; PXL770 500 mg QD: Two capsules were taken BID at least 15 minutes before a meal for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD | Total
Number analyzed (Participants) | 31 | 30 | 30 | 29 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.17) | 52.5 (12.93) | 50.6 (12.26) | 55.7 (12.63) | 52.5 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 23 | 22 | 78
  Male | 15 | 13 | 7 | 7 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 15 | 13 | 7 | 42
  Not Hispanic or Latino | 24 | 15 | 17 | 22 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 2 | 3 | 4 | 10
  White | 27 | 27 | 25 | 24 | 103
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
T2DM status (stratification group) [Count of Participants; unit: Participants]
  T2DM | 14 | 13 | 14 | 12 | 53
  Non-T2DM | 17 | 17 | 16 | 17 | 67

OUTCOME MEASURES:

1. Primary Outcome: Relative Change in the Percentage of Liver Fat Mass (Assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction [MRI-PDFF]) From Baseline to Week 12/End of Treatment (EOT)
Description: MRI acquisitions were performed at pre-qualified local MRI facilities using qualified and standardized instruments at high field strength (3 T or 1.5T) without oral or intravenous contrast. All acquisitions images were transferred to a central reader vendor for central calculation and measurement of MRI-PDFF using the method of Zhong et al. to estimate water and fat components. A 3 cm2 region of interest (ROI) was placed in each Couinaud segment. Central reading was masked to treatment group, clinical data, study site of origin and timepoint.
Time Frame: Baseline to Week 12
Population: Intent-to-treat set (ITTS), defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: percentage
Groups:
- Placebo; PXL770 250 mg QD; PXL770 250 mg BID; PXL770 500 mg QD: Two capsules were taken BID with a glass of water at least 15 minutes before a meal in the morning and in the evening time for 12 weeks
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
percentage | -1.14 (6.344) | -1.03 (6.764) | -14.28 (6.697) | -14.68 (6.452)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.9883, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-15.42 to 15.66], Standard Error of Mean 7.926 — Mean difference (final values) is the difference in Least Squares (LS) Means estimated in the ANCOVA model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.0842, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -13.14, 95% CI 2-sided [-28.06 to 1.78], Standard Error of Mean 7.609 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0763, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -13.54, 95% CI 2-sided [-28.51 to 1.43], Standard Error of Mean 7.636 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model

2. Primary Outcome: Relative Change in the Percentage of Liver Fat Mass (Assessed by MRI-PDFF) From Baseline to Week 12/End of Treatment (Per Protocol Sensitivity Analysis)
Description: MRI acquisitions were performed at pre-qualified local MRI facilities using qualified and standardized instruments at high field strength (3 T or 1.5T) without oral or intravenous contrast. All acquisitions images were transferred to a central reader vendor for central calculation and measurement of MRI-PDFF using the method of Zhong et al. to estimate water and fat components. A 3 cm2 ROI was placed in each Couinaud segment. Central reading was masked to treatment group, clinical data, study site of origin and timepoint.
Time Frame: Baseline to Week 12
Population: Per Protocol Set (PPS), defined as all patients in the ITTS who complete the double-blind treatment period and have an overall treatment duration ≥8 weeks (≥56 days) without any CSR reportable protocol deviations (PD) that is deemed to affect the primary efficacy endpoint of MRI-PDFF.
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 26 | 25 | 23 | 23
percentage | -0.69 (5.818) | -2.27 (6.036) | -13.94 (6.232) | -18.00 (6.012)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.8283, ANCOVA; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-16.01 to 12.85], Standard Error of Mean 7.265 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.0698, ANCOVA; Mean Difference (Final Values) = -13.25, 95% CI 2-sided [-27.60 to 1.10], Standard Error of Mean 7.221 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0184, ANCOVA; Mean Difference (Final Values) = -17.31, 95% CI 2-sided [-31.63 to -2.99], Standard Error of Mean 7.207 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model

3. Primary Outcome: Relative Change in the Percentage of Liver Fat Mass (Assessed by MRI-PDFF) From Baseline to Week 12/End of Treatment (Unstratified Wilcoxon Sensitivity Analysis)
Description: as for outcome 2
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
percentage | 0.49 [-8.68 to 15.46] | 1.44 [-17.85 to 9.31] | -8.32 [-28.91 to 7.29] | -15.29 [-35.87 to 7.06]
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.5537, Wilcoxon (Mann-Whitney); Location Shift = -4.22, 95% CI 2-sided [-15.64 to 8.65]
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.1005, Wilcoxon (Mann-Whitney); Location Shift = -13.64, 95% CI 2-sided [-26.19 to 1.88]
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0387, Wilcoxon (Mann-Whitney); Location Shift = -18.72, 95% CI 2-sided [-31.95 to -1.58]

4. Primary Outcome: Relative Change in the Percentage of Liver Fat Mass (Assessed by MRI-PDFF) From Baseline to Week 12/End of Treatment (Subgroup Analysis - Type 2 Diabetes Mellitus [T2DM])
Description: as for outcome 2
Time Frame: Baseline to Week 12
Population: ITTS T2DM subgroup, defined as all as-randomized T2DM patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 14 | 13 | 14 | 12
percentage | -6.11 (9.745) | 1.15 (9.266) | -16.71 (8.997) | -27.24 (9.572)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.5733, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = 7.25, 95% CI 2-sided [-18.00 to 32.51], Standard Error of Mean 0.5733 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.3861, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -10.61, 95% CI 2-sided [-34.60 to 13.38], Standard Error of Mean 12.236 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.1019, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -21.13, 95% CI 2-sided [-46.46 to 4.19], Standard Error of Mean 12.916 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model

5. Secondary Outcome: Absolute Change in the Percentage of Liver Fat Mass (Assessed by MRI-PDFF) From Baseline to Week 12/End of Treatment
Description: as for outcome 2
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
percentage | 0.023 (1.1117) | -0.218 (1.1801) | -2.548 (1.1988) | -2.391 (1.1399)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.8617, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -0.242, 95% CI 2-sided [-2.961 to 2.478], Standard Error of Mean 1.3873 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.0609, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -2.571, 95% CI 2-sided [-5.260 to 0.117], Standard Error of Mean 1.3712; Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0766, ANCOVA; ANCOVA using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -2.414, 95% CI 2-sided [-5.087 to 0.258], Standard Error of Mean 1.3633 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model

6. Secondary Outcome: Percentage of Responders (Relative Reduction of at Least 30% in Liver Fat Mass) at Week 12/End of Treatment
Description: Responders were defined as patients who achieved a clinically meaningful relative reduction of at least 30% in liver fat mass From baseline to Week 12/EOT as assessed by MRI-PDFF
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
  For patients with missing Week 12/End of Treatment, multiple imputation by fully conditional specification methods was used for analysis, although the n counts and percentages reflect only the observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 27 | 26 | 23 | 24
Participants
  Relative reduction ≥30% | 2 | 4 | 4 | 8
  Relative reduction <30% | 25 | 22 | 19 | 16
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.5592, Regression, Logistic; Logistic regression with multiple imputation; Odds Ratio (OR) = 1.744, 95% CI 2-sided [0.270 to 11.267]
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.3747, Regression, Logistic; Logistic regression with multiple imputation; Odds Ratio (OR) = 2.287, 95% CI 2-sided [0.368 to 14.208]
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0501, Regression, Logistic; Logistic regression with multiple imputation; Odds Ratio (OR) = 5.669, 95% CI 2-sided [1.000 to 32.149]

7. Secondary Outcome: Change in Alanine Amino Transferase (ALT) From Baseline to Week 12/End of Treatment
Description: Blood samples were collected, handled and stored according to the instructions described in the laboratory manual and all measurements were performed at a central laboratory.
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
U/L | 1.0 (2.88) | 0.0 (2.95) | 0.3 (3.10) | -6.3 (3.04)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.8013, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-8.3 to 6.4], Standard Error of Mean 3.71 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.8694, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-8.2 to 7.0], Standard Error of Mean 3.81; Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0581, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-14.9 to 0.3], Standard Error of Mean 3.80; Mean difference (final values) is the difference in LS Means estimated in the MMRM model

8. Secondary Outcome: Change in Aspartate Amino Transferase (AST) From Baseline to Week 12/End of Treatment
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
U/L | -2.8 (1.95) | -1.7 (1.99) | -2.2 (2.08) | -7.0 (2.04)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.6681, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-3.8 to 5.9], Standard Error of Mean 2.44 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.8224, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-4.4 to 5.5], Standard Error of Mean 2.51 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0924, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-9.2 to 0.7], Standard Error of Mean 2.50 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

9. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week12/End of Treatment
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
mmol/L | 0.36 (0.199) | 0.19 (0.205) | -0.17 (0.211) | -0.16 (0.209)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.5148, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.68 to 0.34], Standard Error of Mean 0.256 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.0434, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.05 to -0.02], Standard Error of Mean 0.261 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0494, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.04 to 0.00], Standard Error of Mean 0.261 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

10. Secondary Outcome: Change in Glycated Hemoglobin (HbA1c) From Baseline to Week12/End of Treatment
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
percent | 0.05 (0.092) | -0.08 (0.095) | -0.18 (0.101) | -0.24 (0.096)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.2449, ANCOVA; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.35 to 0.09], Standard Error of Mean 0.111 — Mean difference (final values) is the difference in LS Means estimated in the ANOVA model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.0502, ANCOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.46 to 0.00], Standard Error of Mean 0.115 — Mean difference (final values) is the difference in LS Means estimated in the ANOVA model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0123, ANCOVA; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.51 to -0.06], Standard Error of Mean 0.113 — Mean difference (final values) is the difference in LS Means estimated in the ANOVA model

11. Secondary Outcome: Change in Total Cholesterol From Baseline to Week12/End of Treatment
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
mmol/L | 0.107 (0.1650) | -0.144 (0.1714) | 0.058 (0.1761) | 0.081 (0.1764)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.2510, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.251, 95% CI 2-sided [-0.682 to 0.180], Standard Error of Mean 0.2172 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.8246, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.049, 95% CI 2-sided [-0.486 to 0.388], Standard Error of Mean 0.2202 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.9067, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.026, 95% CI 2-sided [-0.466 to 0.414], Standard Error of Mean 0.2216 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

12. Secondary Outcome: Change in High Density Lipoprotein-Cholesterol (HDL-C) From Baseline to Week12/End of Treatment
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
mmol/L | -0.007 (0.0357) | -0.025 (0.0371) | -0.085 (0.0381) | 0.002 (0.0375)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.6951, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.018, 95% CI 2-sided [-0.111 to 0.075], Standard Error of Mean 0.0468 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.1030, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.078, 95% CI 2-sided [-0.171 to 0.016], Standard Error of Mean 0.0472 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.8583, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.085 to 0.102], Standard Error of Mean 0.0471 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

13. Secondary Outcome: Change in Low Density Lipoprotein-Cholesterol (LDL-C) From Baseline to Week12/End of Treatment
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
mmol/L | 0.011 (0.1401) | -0.094 (0.1391) | 0.155 (0.1427) | 0.092 (0.1456)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.5576, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.105, 95% CI 2-sided [-0.457 to 0.248], Standard Error of Mean 0.1777 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.4261, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.144, 95% CI 2-sided [-0.213 to 0.501], Standard Error of Mean 0.1799 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.6571, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.081, 95% CI 2-sided [-0.281 to 0.443], Standard Error of Mean 0.1822 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

14. Secondary Outcome: Change in Triglycerides From Baseline to Week12/End of Treatment
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
mmol/L | 0.156 (0.2177) | -0.006 (0.2278) | 0.017 (0.2330) | -0.045 (0.2291)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.5732, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.161, 95% CI 2-sided [-0.727 to 0.405], Standard Error of Mean 0.2851 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.6312, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.139, 95% CI 2-sided [-0.712 to 0.434], Standard Error of Mean 0.2884 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.4857, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.201, 95% CI 2-sided [-0.769 to 0.368], Standard Error of Mean 0.2865 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

15. Secondary Outcome: Change in Fibrosis-4 (Fib-4) Score From Baseline to Week 12/End of Treatment
Description: Fib-4 score is a non invasive method based on clinical determinations that indicates the level of fibrosis/ scarring of the liver. The set cutoffs for this scoring are: Fib-4 < 1.45: absence of cirrhosis; Fib-4 between 1.45 - 3.25: inconclusive and Fib-4 > 3.25: cirrhosis.
  Fib-4 score was calculated as (Age [years] × AST [U/L]) / (platelet [10^9/L] × √[ALT [U/L]]). Blood samples used for AST, ALT and platelet counts were collected, handled and stored according to the instructions described in the laboratory manual and all measurements were performed at a central laboratory.
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Fib-4 score
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
Fib-4 score | -0.11 (0.060) | -0.07 (0.062) | -0.09 (0.064) | -0.15 (0.063)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.5737, ANCOVA; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.11 to 0.19], Standard Error of Mean 0.074 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.7563, ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.12 to 0.17], Standard Error of Mean 0.074 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.5695, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.19 to 0.11], Standard Error of Mean 0.075 — Mean difference (final values) is the difference in LS Means estimated in the ANCOVA model

16. Secondary Outcome: Change in Body Weight From Baseline to Week 12/End of Treatment
Description: Body weight was measured using a scale with appropriate resolution, placed on a stable, flat surface. Shoes, bulky layers of clothing, and jackets had to be removed so that only light clothing remained.
Time Frame: Baseline to Week 12
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 31 | 30 | 30 | 29
kg | 0.96 (0.476) | 0.92 (0.486) | 0.20 (0.508) | 0.08 (0.505)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.9552, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-1.34 to 1.27], Standard Error of Mean 0.659 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.2633, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-2.10 to 0.58], Standard Error of Mean 0.674 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.1962, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-2.21 to 0.46], Standard Error of Mean 0.673 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

17. Post Hoc Outcome: Percentage of Responders (Relative Reduction of at Least 30% in Liver Fat Mass) at Week 12/End of Treatment (T2DM Subgroup)
Description: as for outcome 6
Time Frame: Baseline to Week 12
Population: ITTS T2DM subgroup, defined as all as-randomized T2DM patients who received at least one dose of study treatment.
  For patients with missing Week 12/End of Treatment, multiple imputation by fully conditional specification methods was used for analysis, although the n counts and percentages reflect only the observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 11 | 12 | 12 | 10
Participants
  Relative reduction ≥30% | 1 | 2 | 3 | 7
  Relative reduction <30% | 10 | 10 | 9 | 3
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.8245, Regression, Logistic; Odds Ratio (OR) = 1.353, 95% CI 2-sided [0.094 to 19.554]
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.4140, Regression, Logistic; Odds Ratio (OR) = 2.791, 95% CI 2-sided [0.238 to 32.752]
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0341, Regression, Logistic; Odds Ratio (OR) = 14.872, 95% CI 2-sided [1.226 to 180.452]

18. Post Hoc Outcome: Change in ALT From Baseline to Week 12/End of Treatment (T2DM Subgroup)
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS T2DM subgroup, defined as all as-randomized T2DM patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 14 | 13 | 14 | 12
U/L | 2.1 (4.36) | -2.2 (4.20) | -3.8 (4.19) | -12.8 (4.59)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.4626, Mixed Models Analysis; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-16.1 to 7.5], Standard Error of Mean 5.84 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.3160, Mixed Models Analysis; Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-17.9 to 5.9], Standard Error of Mean 5.88 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0204, Mixed Models Analysis; Mean Difference (Final Values) = -14.9, 95% CI 2-sided [-27.4 to -2.4], Standard Error of Mean 6.19 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

19. Post Hoc Outcome: Change in AST From Baseline to Week 12/End of Treatment (T2DM Subgroup)
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS T2DM subgroup, defined as all as-randomized T2DM patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 14 | 13 | 14 | 12
U/L | -0.8 (2.92) | -3.7 (2.87) | -0.9 (2.82) | -10.7 (3.09)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.4601, Mixed Models Analysis; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-10.8 to 5.0], Standard Error of Mean 3.91 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.9782, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-8.1 to 7.9], Standard Error of Mean 3.95 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0205, Mixed Models Analysis; Mean Difference (Final Values) = -9.9, 95% CI 2-sided [-18.3 to -1.6], Standard Error of Mean 4.13 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

20. Post Hoc Outcome: Change in FPG From Baseline to Week12/End of Treatment (T2DM Subgroup)
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS T2DM subgroup, defined as all as-randomized T2DM patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 14 | 13 | 14 | 12
mmol/L | 0.54 (0.399) | 0.51 (0.404) | -0.29 (0.384) | -0.65 (0.427)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.9529, Mixed Models Analysis; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-1.12 to 1.05], Standard Error of Mean 0.538 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.1285, Mixed Models Analysis; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.90 to 0.25], Standard Error of Mean 0.532 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0417, Mixed Models Analysis; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-2.32 to -0.05], Standard Error of Mean 0.565 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

21. Post Hoc Outcome: Change in HbA1c From Baseline to Week12/End of Treatment (T2DM Subgroup)
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: ITTS T2DM subgroup, defined as all as-randomized T2DM patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
Number analyzed (Participants) | 14 | 13 | 14 | 12
percent | 0.20 (0.175) | -0.04 (0.176) | -0.23 (0.175) | -0.44 (0.188)
Statistical Analysis 1: Comparison: Placebo vs PXL770 250 mg QD; Test type: Superiority; p = 0.3141, ANCOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.69 to 0.23], Standard Error of Mean 0.228 — Mean difference (final values) is the difference in LS Means estimated in the ANOVA model
Statistical Analysis 2: Comparison: Placebo vs PXL770 250 mg BID; Test type: Superiority; p = 0.0656, ANCOVA; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.88 to 0.03], Standard Error of Mean 0.226 — Mean difference (final values) is the difference in LS Means estimated in the ANOVA model
Statistical Analysis 3: Comparison: Placebo vs PXL770 500 mg QD; Test type: Superiority; p = 0.0101, ANCOVA; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.12 to -0.16], Standard Error of Mean 0.237 — Mean difference (final values) is the difference in LS Means estimated in the ANOVA model

ADVERSE EVENTS:
Time Frame: All AEs were collected from the time of ICF signature to the End-of-study Visit, ie 19 weeks on average. Only events that occur after the first dose intake of IMP of the Double-blind (DB) treatment period or if they were present prior to the first intake of IMP of the DB treatment period and increased in severity or relationship to IMP after the first intake of IMP of the DB treatment period were considered as Treatment Emergent Adverse Events (TEAEs). Only TEAEs are presented in this section.
Arm/Group | Placebo | PXL770 250 mg QD | PXL770 250 mg BID | PXL770 500 mg QD
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 2/30 | 1/29
Other Adverse Events (participants affected / at risk) | 8/31 | 13/30 | 14/30 | 13/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | PXL770 250 mg QD (N=30) | PXL770 250 mg BID (N=30) | PXL770 500 mg QD (N=29)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | PXL770 250 mg QD (N=30) | PXL770 250 mg BID (N=30) | PXL770 500 mg QD (N=29)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 7 (8) | 6 (7)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (6) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 4 (5) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT03763877/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT03763877/SAP_001.pdf